CLINICAL TRIAL: NCT00069004
Title: Prevalence of Morphologic and Metabolic Abnormalities in Vertically HIV-Infected and Uninfected Children and Youth
Brief Title: A Study of Physical and Metabolic Abnormalities in HIV Infected and Uninfected Children and Youth
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: P1045; 10108 (Registry Identifier: DAIDS ES); PACTG P1045
Record Dates: First submitted 2003-09-12; First posted 2003-09-16 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: HIV Infections; HIV-Associated Lipodystrophy Syndrome; HIV Lipodystrophy Syndrome; Lipodystrophy; Dyslipidemia; Osteoporosis; Osteopenia
Keywords: HIV-Associated Lipodystrophy Syndrome; HIV Lipodystrophy Syndrome; Treatment Experienced; Lipodystrophy; Dyslipidemia; Osteoporosis; Osteopenia
MeSH Terms: conditions — HIV Infections; HIV-Associated Lipodystrophy Syndrome; Lipodystrophy; Dyslipidemias; Osteoporosis; Bone Diseases, Metabolic

SUMMARY:
The purpose of this study is to assess the prevalence of metabolic and physical abnormalities in HIV infected (via mother-to-child transmission) and uninfected children and youth. Metabolism, body composition, bone density, and other factors will be assessed in relationship to participants' exposure to highly active antiretroviral therapy (HAART).

DETAILED DESCRIPTION:
Despite advances in HIV care associated with HAART, many patients on HAART regimens develop physical and metabolic problems, including changes in body fat distribution (lipodystrophy), osteopenia and osteoporosis, dyslipidemia, and hyperlactatemia. Early studies suggest that protease inhibitors (PIs) were directly responsible for HIV Lipodystrophy Syndrome (HLS) and skeletal complications in HAART-treated patients. This study will compare HIV infected, HAART-treated children and youth and their uninfected counterparts to make connections between HAART, HLS, and skeletal and metabolic problems. The study is the first to address the prevalence and risk assessment of these complications in children, and will be useful in predicting long-term prognosis in HIV patients who use or have used HAART.

There will be three groups in the study. Group 1 participants will be uninfected volunteers who will receive no protocol-specific treatment or other intervention. Vertically infected HIV patients in Groups 2 and 3 will continue their current HAART either on a non-PI-containing regimen (Group 2) or a PI-containing regimen (Group 3). Screening evaluations will be conducted within 30 days prior to study entry. Study evaluations may be completed at study entry or over the course of up to 3 study visits. All participants will undergo whole body and regional DEXA scans (to assess bone density), measurements to determine sexual maturity, and blood work.

ELIGIBILITY:
Inclusion Criteria

For HIV uninfected participants (Group 1)

* HIV-1 negative (perinatally HIV-exposed but uninfected participants are eligible)

For HIV infected participants (Groups 2 and 3)

* Mother-to-child (vertically) transmitted HIV infection
* Confirmed diagnosis of HIV-1 infection by two positive assays from two different samples
* For Group 2, cannot have taken a PI-containing regimen in the 12 months prior to study entry or have ever received a PI for 2 or more weeks
* For Group 3, must currently be taking the same PI-containing regimen taken continuously for at least 12 months prior to study entry

For all participants

* Accessible medical and medications history
* Parent, legal guardian, or participant willing to give informed consent and willing to comply with study requirements
* Females who have begun menstruating must have negative pregnancy test

Exclusion Criteria

* Receipt of certain medications, including growth hormone, megestrol acetate, anabolic agents, anticytokine agents, systemic ketoconazole, systemic glucocorticoids (except if receiving stable physiologic doses), or drugs to treat osteoporosis
* Type II diabetes mellitus and unable to omit medication prior to specimen collection
* Pregnancy within the last 12 months, currently pregnant, or breastfeeding
* History of eating disorder

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 450
Dates: Start 2003-10; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace Aldrovandi, MD, Study Chair — University of Alabama at Birmingham; Peggy Borum, PhD, Study Chair — University of Florida
Locations (38):
- United States (36):
  - UAB, Dept. of Ped., Div. of Infectious Diseases, Birmingham, Alabama
  - Usc La Nichd Crs, Alhambra, California
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - UCSD Mother-Child-Adolescent Program CRS, San Diego, California
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Harbor - UCLA Med. Ctr. - Dept. of Peds., Div. of Infectious Diseases, Torrance, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Yale Univ. School of Medicine - Dept. of Peds., Div. of Infectious Disease, New Haven, Connecticut
  - Children's National Med. Ctr., ACTU, Washington D.C., District of Columbia
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - South Florida CDTC Ft Lauderdale NICHD CRS, Fort Lauderdale, Florida
  - Univ. of Florida College of Medicine-Dept of Peds, Div. of Immunology, Infectious Diseases & Allergy, Gainesville, Florida
  - USF - Tampa NICHD CRS, Tampa, Florida
  - Med. College of Georgia School of Medicine, Dept. of Peds., Div. of Infectious Diseases, Augusta, Georgia
  - Mt. Sinai Hosp. Med. Ctr. - Chicago, Womens & Childrens HIV Program, Chicago, Illinois
  - Chicago Children's CRS, Chicago, Illinois
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Johns Hopkins Hosp. & Health System - Dept. of Peds., Div. of Infectious Diseases, Baltimore, Maryland
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - UMDNJ - Robert Wood Johnson Med. School, Div. of Allergy, Immunology & Infectious Diseases, New Brunswick, New Jersey
  - Rutgers - New Jersey Medical School CRS, Newark, New Jersey
  - SUNY Downstate Med. Ctr., Children's Hosp. at Downstate NICHD CRS, Brooklyn, New York
  - Nyu Ny Nichd Crs, New York, New York
  - Metropolitan Hosp. Ctr., New York, New York
  - Mt. Sinai School of Medicine, Div. of Ped. Infectious Diseases, New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - Strong Memorial Hospital Rochester NY NICHD CRS, Rochester, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - Lincoln Med. & Mental Health Ctr., The Bronx, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - Jacobi Med. Ctr., The Bronx, New York
  - UNC at Chapel Hill School of Medicine - Dept. of Peds., Div. of Immunology & Infectious Diseases, Chapel Hill, North Carolina
  - DUMC Ped. CRS, Durham, North Carolina
  - St. Jude/UTHSC CRS, Memphis, Tennessee
  - Texas Children's Hosp. CRS, Houston, Texas
- Puerto Rico (2):
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan

REFERENCES:
- [Background] Wanke CA, Falutz JM, Shevitz A, Phair JP, Kotler DP. Clinical evaluation and management of metabolic and morphologic abnormalities associated with human immunodeficiency virus. Clin Infect Dis. 2002 Jan 15;34(2):248-59. doi: 10.1086/324744. Epub 2001 Dec 7. PMID 11740715
- [Background] Smith KY. Selected metabolic and morphologic complications associated with highly active antiretroviral therapy. J Infect Dis. 2002 May 15;185 Suppl 2:S123-7. doi: 10.1086/340200. PMID 12001033
- [Background] Currier J, Carpenter C, Daar E, Kotler D, Wanke C. Identifying and managing morphologic complications of HIV and HAART. AIDS Read. 2002 Mar;12(3):114-9, 124-5. PMID 11966241
- [Background] Carr A, Samaras K, Thorisdottir A, Kaufmann GR, Chisholm DJ, Cooper DA. Diagnosis, prediction, and natural course of HIV-1 protease-inhibitor-associated lipodystrophy, hyperlipidaemia, and diabetes mellitus: a cohort study. Lancet. 1999 Jun 19;353(9170):2093-9. doi: 10.1016/S0140-6736(98)08468-2. PMID 10382692
- [Background] Bockhorst JL, Ksseiry I, Toye M, Chipkin SR, Stechenberg BW, Fisher DJ, Allen HF. Evidence of human immunodeficiency virus-associated lipodystrophy syndrome in children treated with protease inhibitors. Pediatr Infect Dis J. 2003 May;22(5):463-5. PMID 12797313
- [Background] Tebas P, Powderly WG, Claxton S, Marin D, Tantisiriwat W, Teitelbaum SL, Yarasheski KE. Accelerated bone mineral loss in HIV-infected patients receiving potent antiretroviral therapy. AIDS. 2000 Mar 10;14(4):F63-7. doi: 10.1097/00002030-200003100-00005. PMID 10770534
- [Result] Jacobson DL, Lindsey JC, Gordon CM, Moye J, Hardin DS, Mulligan K, Aldrovandi GM; Pediatric AIDS Clinical Trials Group P1045 team. Total body and spinal bone mineral density across Tanner stage in perinatally HIV-infected and uninfected children and youth in PACTG 1045. AIDS. 2010 Mar 13;24(5):687-96. doi: 10.1097/QAD.0b013e328336095d. PMID 20168204